CLINICAL TRIAL: NCT01466868
Title: A Phase II Study of MK 2206 in Patients With Relapsed or Refractory Diffuse Large B Cell Lymphoma
Brief Title: Study of MK 2206 in Patients With Relapsed or Refractory Diffuse Large B Cell Lymphoma
Acronym: AKTIL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Regarding the comments of the iDSMB, the sponsor decided to stop the inclusions
Sponsor: Centre Leon Berard (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AKTIL
Record Dates: First submitted 2011-10-28; First posted 2011-11-08 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Diffuse Large B cell Lymphoma; AKT; MK 2206; objective response rate; progression free survival; overall survival; safety
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — MK 2206

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MK2206 (Experimental): Treatment is started the day after registration (day 1)until progression according to Cheson international response criteria or documented toxicity.
  Interventions: Drug: MK2206

INTERVENTIONS:
Drug: MK2206 — Treatment will be administered orally once weekly, 2 hours before or after a meal, at day 1, 8, 15, 22 over a 28 day cycle period.
  The starting dose level is 200 mg. 2 dose reduction are allowed (135 mg and 90 mg)in case of documented toxicity according to the specific algorithms.

SUMMARY:
The purpose of this study is to evaluate the antitumor efficacy and the safety of MK 2206 in patients with relapsed or refractory diffuse large B cell lymphoma.

DETAILED DESCRIPTION:
Diffuse Large B-cell Lymphoma (DLBCL) is the most frequent subtype of Non-Hodgkin lymphoma (NHL) around the world, in all age groups.

DLBCL is a curable disease and combination of monoclonal antibody against CD20 (rituximab) with cyclophosphamide, doxorubicin, vincristine and prednisolone (CHOP) regimen have improved the prognosis of patients with a 20% increase of the cure rate. For the remaining patients who are not in complete response and/or who relapse after first line therapy, the possibility of cure is dramatically reduced.

As PI3K/AKT/mTOR pathway regulates the expression of cyclin D1, c-Myc and Stat3 proteins, which are involved in the pathogenesis of DLBCL HL), this signalling axis is an emerging therapeutic target for treatment of DLBCL.

One study has shown that the level of p-Akt is an adverse prognostic feature in DLBCL and is found in 52% of tumors samples from DLBCL patients.

Given the fact that AKT is overactivated in about to 52% of DLBCL and is considered as a poor prognosis factor, we postulate that targeting AKT in DLBCL may be an interesting therapeutic strategy.

MK-2206 is an orally selective allosteric inhibitor of AKT developed by MERCK currently highlighted as a promising therapeutic option for cancer patients and under clinical development in several Phase 1 trials.

Therefore, we propose to conduct a Phase II study using a two-stage Simon's design with objective response rate (ORR) as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diffuse large B-Cell lymphomas.
* Patients must have measurable disease.
* Subjects must have received at least two prior treatment lines.There is no maximal limit on the number of prior therapies

  * Prior treatment must include CHOP (cyclophosphamide, doxorubicin, vincristine and prednisolone) -like chemotherapy in combination with rituximab. Rituximab used alone is not considered as a separate regimen.
  * Prior treatment could include high dose chemotherapy with autologous stem-cell transplantation if patients had progressed ≥ 3 months after this treatment.
  * Salvage treatment, mobilization chemotherapy, high-dose chemotherapy and planned post-transplant therapy should be considered as one regimen
  * Relapsed or refractory patients who are candidate to high-dose chemotherapy and autologous or allogenic stem cell transplantation are not eligible.
* Patients must have discontinued all prior therapies for at least 5 times the t1/2 of prior anti-cancer therapies before study entry.
* Male or female patients, age ≥ 18 years.
* Life expectancy greater than 4 months.
* ECOG performance status ≤2.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1.5 x 109/L,
  * Platelet count ≥ 100 x 109/L or ≥75 x 109/L if the bone marrow is involved,
  * AST/ALT ≤ 2.5 x upper limit of normal (ULN) (or ≤ 5.0 x ULN if liver metastasis) direct bilirubin ≤ 1.5ULN
  * Calculated creatinine clearance (Cockcroft-Gault formula) of ≥ 50mL/min
* Patients must agree to use adequate double contraception
* Patients must be able to swallow whole tablets.
* Cardiovascular baseline QTcF≤ 450 msec (male) or QTcF≤470msec (female).
* Signed written informed consent document.
* Patients with French Social Security in compliance with the French law relating to biomedical research.

Exclusion Criteria:

* Tumor tissue sample not available for pathological review.
* Patients with others than Diffuse large B-Cell Lymphoma histology.
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
* Patients who have not recovered from adverse events grade > 1 due to agents administered more than 4 weeks earlier.
* Patients who are receiving any other investigational agents.
* Patients with known CNS involvement should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the compliance to the study protocol.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-2206 tablets.
* Patients with uncontrolled hyperglycemia
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and breastfeeding women are excluded from this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with MK-2206.
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption.
* Patients with clinically important history of liver disease, including viral or other hepatitis or cirrhosis.
* Prior history of malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for ≥ 3 years.
* Uncontrolled hypertension with resting SBP>140 or resting DBP>90mm Hg

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-11; Primary Completion 2013-09 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
evaluation of the antitumor activity of MK-2206 in terms of objective response rate (ORR). | 4 months after the first day of treatment.
  the objective response rate (ORR) is measured as per 2007 Cheson international response criteria.

SECONDARY OUTCOMES:
safety profile | during the treatment and up to 3.5 years from the first inclusion
  safety profile is characterized by type, frequency and seriousness of the toxicities showed by patients and graded using CTCAE-V04.
overall survival | from the date of inclusion to the date of death from any cause (up to 3.5 years from the first inclusion)
progression-free survival | from the date of inclusion to the date of event defined as the first documented disease progression or death from any cause (up to 3.5 years from the first inclusion)
duration of response | from the time of first documented response (complete response or partial response) until the first documented disease progression or death due to underlying cancer (up to 3.5 years from the first inclusion)
evaluation of the antitumor activity of MK-2206 in terms of objective response rate (ORR). | 4 months after the first day of treatment
  the objective response rate (ORR) is measured as per 1999 Cheson international response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Ghesquières, MD, Principal Investigator — Centre Leon Berard, Lyon, France; Philippe Cassier, MD, Principal Investigator — Centre Leon Berard
Locations (13):
- France (13):
  - Institut Bergonié, Bordeaux
  - Centre Henri Mondor, Créteil
  - CHRU, Lille
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHU St Eloi, Montpellier
  - CHU, Nancy
  - CHU de Nantes, Nantes
  - Hôpital Saint-Louis, Paris
  - Hôpital Necker, Paris
  - Centre Hospitalier LYON SUD, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Thieblemont C, Gisselbrecht C. Second-line treatment paradigms for diffuse large B-cell lymphomas. Curr Oncol Rep. 2009 Sep;11(5):386-93. doi: 10.1007/s11912-009-0052-0. PMID 19679014
- [Background] Philip T, Guglielmi C, Hagenbeek A, Somers R, Van der Lelie H, Bron D, Sonneveld P, Gisselbrecht C, Cahn JY, Harousseau JL, et al. Autologous bone marrow transplantation as compared with salvage chemotherapy in relapses of chemotherapy-sensitive non-Hodgkin's lymphoma. N Engl J Med. 1995 Dec 7;333(23):1540-5. doi: 10.1056/NEJM199512073332305. PMID 7477169
- [Background] Gisselbrecht C, Glass B, Mounier N, Singh Gill D, Linch DC, Trneny M, Bosly A, Ketterer N, Shpilberg O, Hagberg H, Ma D, Briere J, Moskowitz CH, Schmitz N. Salvage regimens with autologous transplantation for relapsed large B-cell lymphoma in the rituximab era. J Clin Oncol. 2010 Sep 20;28(27):4184-90. doi: 10.1200/JCO.2010.28.1618. Epub 2010 Jul 26. PMID 20660832
- [Background] Feugier P, Van Hoof A, Sebban C, Solal-Celigny P, Bouabdallah R, Ferme C, Christian B, Lepage E, Tilly H, Morschhauser F, Gaulard P, Salles G, Bosly A, Gisselbrecht C, Reyes F, Coiffier B. Long-term results of the R-CHOP study in the treatment of elderly patients with diffuse large B-cell lymphoma: a study by the Groupe d'Etude des Lymphomes de l'Adulte. J Clin Oncol. 2005 Jun 20;23(18):4117-26. doi: 10.1200/JCO.2005.09.131. Epub 2005 May 2. PMID 15867204
- [Background] Lignon J, Sibon D, Madelaine I, Brice P, Franchi P, Briere J, Mounier N, Gisselbrecht C, Faure P, Thieblemont C. Rituximab, dexamethasone, cytarabine, and oxaliplatin (R-DHAX) is an effective and safe salvage regimen in relapsed/refractory B-cell non-Hodgkin lymphoma. Clin Lymphoma Myeloma Leuk. 2010 Aug;10(4):262-9. doi: 10.3816/CLML.2010.n.055. PMID 20709662
- [Background] Coiffier B. Fourteen years of high-dose CHOP (ACVB regimen): preliminary conclusions about the treatment of aggressive-lymphoma patients. Hamilton Fairley Award Lecture, European Society for Medical Oncology Meeting, Lisbon, November 21, 1994. Ann Oncol. 1995 Mar;6(3):211-7. doi: 10.1093/oxfordjournals.annonc.a059149. No abstract available. PMID 7612487
- [Background] Wilson WH, Dunleavy K, Pittaluga S, Hegde U, Grant N, Steinberg SM, Raffeld M, Gutierrez M, Chabner BA, Staudt L, Jaffe ES, Janik JE. Phase II study of dose-adjusted EPOCH and rituximab in untreated diffuse large B-cell lymphoma with analysis of germinal center and post-germinal center biomarkers. J Clin Oncol. 2008 Jun 1;26(16):2717-24. doi: 10.1200/JCO.2007.13.1391. Epub 2008 Mar 31. PMID 18378569
- [Background] Dupuis J, Itti E, Rahmouni A, Hemery F, Gisselbrecht C, Lin C, Copie-Bergman C, Belhadj K, El Gnaoui T, Gaillard I, Kuhnowski F, Meignan M, Haioun C. Response assessment after an inductive CHOP or CHOP-like regimen with or without rituximab in 103 patients with diffuse large B-cell lymphoma: integrating 18fluorodeoxyglucose positron emission tomography to the International Workshop Criteria. Ann Oncol. 2009 Mar;20(3):503-7. doi: 10.1093/annonc/mdn671. Epub 2008 Dec 11. PMID 19074215
- [Background] Shipp MA. Molecular signatures define new rational treatment targets in large B-cell lymphomas. Hematology Am Soc Hematol Educ Program. 2007:265-9. doi: 10.1182/asheducation-2007.1.265. PMID 18024639
- [Background] Altomare DA, Testa JR. Perturbations of the AKT signaling pathway in human cancer. Oncogene. 2005 Nov 14;24(50):7455-64. doi: 10.1038/sj.onc.1209085. PMID 16288292
- [Background] Hennessy BT, Smith DL, Ram PT, Lu Y, Mills GB. Exploiting the PI3K/AKT pathway for cancer drug discovery. Nat Rev Drug Discov. 2005 Dec;4(12):988-1004. doi: 10.1038/nrd1902. PMID 16341064
- [Background] Steelman LS, Stadelman KM, Chappell WH, Horn S, Basecke J, Cervello M, Nicoletti F, Libra M, Stivala F, Martelli AM, McCubrey JA. Akt as a therapeutic target in cancer. Expert Opin Ther Targets. 2008 Sep;12(9):1139-65. doi: 10.1517/14728222.12.9.1139. PMID 18694380
- [Background] Sarbassov DD, Ali SM, Sabatini DM. Growing roles for the mTOR pathway. Curr Opin Cell Biol. 2005 Dec;17(6):596-603. doi: 10.1016/j.ceb.2005.09.009. Epub 2005 Oct 13. PMID 16226444
- [Background] Gupta M, Ansell SM, Novak AJ, Kumar S, Kaufmann SH, Witzig TE. Inhibition of histone deacetylase overcomes rapamycin-mediated resistance in diffuse large B-cell lymphoma by inhibiting Akt signaling through mTORC2. Blood. 2009 Oct 1;114(14):2926-35. doi: 10.1182/blood-2009-05-220889. Epub 2009 Jul 29. PMID 19641186
- [Background] Hay N. The Akt-mTOR tango and its relevance to cancer. Cancer Cell. 2005 Sep;8(3):179-83. doi: 10.1016/j.ccr.2005.08.008. PMID 16169463
- [Background] Weil RJ. Incorporating molecular tools into early-stage clinical trials. PLoS Med. 2008 Jan 22;5(1):e21. doi: 10.1371/journal.pmed.0050021. PMID 18215108
- [Background] Kawauchi K, Ogasawara T, Yasuyama M, Otsuka K, Yamada O. The PI3K/Akt pathway as a target in the treatment of hematologic malignancies. Anticancer Agents Med Chem. 2009 Jun;9(5):550-9. doi: 10.2174/187152009788451851. PMID 19519296
- [Background] Testa JR, Bellacosa A. AKT plays a central role in tumorigenesis. Proc Natl Acad Sci U S A. 2001 Sep 25;98(20):10983-5. doi: 10.1073/pnas.211430998. No abstract available. PMID 11572954
- [Background] Hasselblom S, Hansson U, Olsson M, Toren L, Bergstrom A, Nilsson-Ehle H, Andersson PO. High immunohistochemical expression of p-AKT predicts inferior survival in patients with diffuse large B-cell lymphoma treated with immunochemotherapy. Br J Haematol. 2010 May;149(4):560-8. doi: 10.1111/j.1365-2141.2010.08123.x. Epub 2010 Mar 1. PMID 20201946
- [Background] Uddin S, Hussain AR, Siraj AK, Manogaran PS, Al-Jomah NA, Moorji A, Atizado V, Al-Dayel F, Belgaumi A, El-Solh H, Ezzat A, Bavi P, Al-Kuraya KS. Role of phosphatidylinositol 3'-kinase/AKT pathway in diffuse large B-cell lymphoma survival. Blood. 2006 Dec 15;108(13):4178-86. doi: 10.1182/blood-2006-04-016907. Epub 2006 Aug 31. PMID 16946303
- [Background] Wanner K, Hipp S, Oelsner M, Ringshausen I, Bogner C, Peschel C, Decker T. Mammalian target of rapamycin inhibition induces cell cycle arrest in diffuse large B cell lymphoma (DLBCL) cells and sensitises DLBCL cells to rituximab. Br J Haematol. 2006 Sep;134(5):475-84. doi: 10.1111/j.1365-2141.2006.06210.x. PMID 16856892
- [Background] Reeder CB, Gornet MK, Habermann TM, et al.: A phase II trial of the oral mTOR inhibitor Everolimus (RAD001) in relapsed aggressive Non-Hodgkin Lymphoma (NHL), in (ed 110; Abstract 121), 2007
- [Background] Johnson PB, Ansell SM, Colgan JP, et al.: Phase II trial of the oral mTOR inhibitor everolimus (RAD001) for patients with relapsed or refractory lymphoma, in (ed 25, No. 18S, Abstract 8055), 2007
- [Background] Smith SM, van Besien K, Karrison T, Dancey J, McLaughlin P, Younes A, Smith S, Stiff P, Lester E, Modi S, Doyle LA, Vokes EE, Pro B. Temsirolimus has activity in non-mantle cell non-Hodgkin's lymphoma subtypes: The University of Chicago phase II consortium. J Clin Oncol. 2010 Nov 1;28(31):4740-6. doi: 10.1200/JCO.2010.29.2813. Epub 2010 Sep 13. PMID 20837940
- [Background] Woehrer S, Hejna M, Skrabs C, Drach J, Zielinski CC, Jaeger U, Raderer M. Rituximab, Ara-C, dexamethasone and oxaliplatin is safe and active in heavily pretreated patients with diffuse large B-cell lymphoma. Oncology. 2005;69(6):499-502. doi: 10.1159/000091031. Epub 2006 Jan 16. PMID 16424679
- [Background] Wiernik PH, Lossos IS, Tuscano JM, Justice G, Vose JM, Cole CE, Lam W, McBride K, Wride K, Pietronigro D, Takeshita K, Ervin-Haynes A, Zeldis JB, Habermann TM. Lenalidomide monotherapy in relapsed or refractory aggressive non-Hodgkin's lymphoma. J Clin Oncol. 2008 Oct 20;26(30):4952-7. doi: 10.1200/JCO.2007.15.3429. Epub 2008 Jul 7. PMID 18606983
- [Background] Goy A, Younes A, McLaughlin P, Pro B, Romaguera JE, Hagemeister F, Fayad L, Dang NH, Samaniego F, Wang M, Broglio K, Samuels B, Gilles F, Sarris AH, Hart S, Trehu E, Schenkein D, Cabanillas F, Rodriguez AM. Phase II study of proteasome inhibitor bortezomib in relapsed or refractory B-cell non-Hodgkin's lymphoma. J Clin Oncol. 2005 Feb 1;23(4):667-75. doi: 10.1200/JCO.2005.03.108. Epub 2004 Dec 21. PMID 15613697
- [Background] Robertson MJ, Kahl BS, Vose JM, de Vos S, Laughlin M, Flynn PJ, Rowland K, Cruz JC, Goldberg SL, Musib L, Darstein C, Enas N, Kutok JL, Aster JC, Neuberg D, Savage KJ, LaCasce A, Thornton D, Slapak CA, Shipp MA. Phase II study of enzastaurin, a protein kinase C beta inhibitor, in patients with relapsed or refractory diffuse large B-cell lymphoma. J Clin Oncol. 2007 May 1;25(13):1741-6. doi: 10.1200/JCO.2006.09.3146. Epub 2007 Mar 26. PMID 17389337
- [Background] Casasnovas RO, Meignan M, Berriolo-Riedinger A, Bardet S, Julian A, Thieblemont C, Vera P, Bologna S, Briere J, Jais JP, Haioun C, Coiffier B, Morschhauser F; Groupe d'etude des lymphomes de l'adulte (GELA). SUVmax reduction improves early prognosis value of interim positron emission tomography scans in diffuse large B-cell lymphoma. Blood. 2011 Jul 7;118(1):37-43. doi: 10.1182/blood-2010-12-327767. Epub 2011 Apr 25. PMID 21518924
- [Background] Juweid ME, Stroobants S, Hoekstra OS, Mottaghy FM, Dietlein M, Guermazi A, Wiseman GA, Kostakoglu L, Scheidhauer K, Buck A, Naumann R, Spaepen K, Hicks RJ, Weber WA, Reske SN, Schwaiger M, Schwartz LH, Zijlstra JM, Siegel BA, Cheson BD; Imaging Subcommittee of International Harmonization Project in Lymphoma. Use of positron emission tomography for response assessment of lymphoma: consensus of the Imaging Subcommittee of International Harmonization Project in Lymphoma. J Clin Oncol. 2007 Feb 10;25(5):571-8. doi: 10.1200/JCO.2006.08.2305. Epub 2007 Jan 22. PMID 17242397
- [Background] Cheson BD, Horning SJ, Coiffier B, Shipp MA, Fisher RI, Connors JM, Lister TA, Vose J, Grillo-Lopez A, Hagenbeek A, Cabanillas F, Klippensten D, Hiddemann W, Castellino R, Harris NL, Armitage JO, Carter W, Hoppe R, Canellos GP. Report of an international workshop to standardize response criteria for non-Hodgkin's lymphomas. NCI Sponsored International Working Group. J Clin Oncol. 1999 Apr;17(4):1244. doi: 10.1200/JCO.1999.17.4.1244. PMID 10561185
- [Background] Meignan M, Itti E, Gallamini A, Haioun C. Interim 18F-fluorodeoxyglucose positron emission tomography in diffuse large B-cell lymphoma: qualitative or quantitative interpretation--where do we stand? Leuk Lymphoma. 2009 Nov;50(11):1753-6. doi: 10.3109/10428190903308056. PMID 19863178
- [Background] Meignan M, Gallamini A, Haioun C, Polliack A. Report on the Second International Workshop on interim positron emission tomography in lymphoma held in Menton, France, 8-9 April 2010. Leuk Lymphoma. 2010 Dec;51(12):2171-80. doi: 10.3109/10428194.2010.529208. Epub 2010 Nov 15. PMID 21077737